CLINICAL TRIAL: NCT00118586
Title: Neuropathological Basis of Spasmodic Dysphonia and Related Voice Disorders
Brief Title: Neuropathology of Spasmodic Dysphonia
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050189; 05-N-0189
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Voice Disorders; Spasmodic Dysphonia; Healthy; Movement Disorder; Focal Dystonia
Keywords: Neuroanatomy; Brain Damage; Dystonia; Pathology; Brain Imaging; Natural History; Spasmodic Dysphonia; SD; Focal Dystonia; Healthy Volunteer; HV
MeSH Terms: conditions — Voice Disorders; Dysphonia; Movement Disorders; Dystonic Disorders; Brain Injuries; Dystonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Muscle tension dysphonia: Increased phonatory muscle tension in the paralaryngeal and suprahyoid muscles onpalpation
- Normal Volunteers: Normal vocal function refers to normal voice quality with a negative history of voice orlaryngeal disorders
- Spasmodic dysphonia: A diagnosis of adductor or abductor SD will be based on voice testing and fiberoptic nasolaryngoscopy conducted during the initial interview
- Vocal Tremor: Vocal tremor during vocalization that primarily involves laryngeal structures

SUMMARY:
This study will look for abnormalities in a brain of persons affected with spasmodic dysphonia, a form of movement disorder that involves involuntary "spasms" of the muscles in the vocal folds causing breaks of speech and affecting voice quality. The causes of this disorder are not known. The study will compare results of magnetic resonance imaging (MRI) in people with spasmodic dysphonia and in healthy volunteers.

People with adductor or abductor spasmodic dysphonia and healthy volunteers may be eligible for this study. Candidates are screened with a medical history, physical examination, and a test called nasolaryngoscopy. For this test, the inside of the subject's nose is sprayed with a decongestant, and a small, flexible tube called a nasolaryngoscope is passed through the nose to the back of the throat to allow examination of the larynx (voice box). During this procedure, the subject is asked to perform tasks such as talking, singing, whistling, and saying prolonged vowels. The nasolaryngoscope is connected to a camera to record the movements of the vocal folds during these tasks.

Eligible participants then undergo MRI of the brain. MRI uses a strong magnetic field and radio waves instead of x-rays to obtain images of body organs and tissues. For this test, the subject lies on a table that slides into the MRI scanner, a narrow metal cylinder, wearing ear plugs to muffle loud knocking sound that occurs during the scan. During MRI anatomical images of the brain are obtained. Subject may be asked to participate in up to two scanning sessions. Each session takes about 1-1/2 hours.

Participants may also be asked to volunteer for a brain donation program which is optional. Information gained from donated tissue may lead to better treatments and potential cures for spasmodic dysphonia.

DETAILED DESCRIPTION:
Spasmodic dysphonia (SD) is a focal dystonia affecting the neural control of the laryngeal musculature for speech production. Although the clinical symptoms of SD have been described, the underlying pathological mechanisms remain unknown. Treatment strategies are of short benefit and expensive.

Muscle tension dysphonia (MTD) is considered a behavioral voice disorder because many cases benefit from behavioral therapy. The etiology of this vocal misuse disorder remains unknown but is not considered neurological and is thought to differ from SD.

Vocal tremor (VT) is a form of benign essential tremor. In less severely affected persons, vocal tremor is action-induced and occurs during vocalization only. In more severe cases, the tremor can be present also during exhalation and whispering and affect other structures, such as the velum and pharynx. This is also considered a neurological disorder but may differ in character from SD. Both these disorders can co-occur with SD but can also occur independently.

The anatomical characteristics of pre- and postmortem brains in patients with SD, MTD and VT and healthy volunteers will be investigated using imaging and neurohistological techniques to provide insight into the pathogenesis of SD. Identification of the neuropathological basis of SD and how it differs from other voice disorders would enhance our understanding of the neurological basis of SD.

OBJECTIVES:

Our objective in this study is to investigate anatomical and morphological characteristics of premortem and postmortem brains from persons with SD, and determine how it differs from other voice disorders such as MTD and VT using magnetic resonance imaging (MRI), diffusion tensor imaging (DTI), and neurohistological techniques.

STUDY POPULATION:

We plan to examine persons referred with a diagnosis of SD, MTD, and VT to confirm whether they have symptoms of the disorder and to identify research volunteers who are without neurological, psychiatric, or head and neck disorders. The research volunteers could be spouses of persons with SD, MTD, and VT without a familial relationship.

DESIGN:

This is a natural history study. In the premortem part of the study persons with SD, MTD, and VT and research volunteers will be screened for eligibility for the study. Brain MRI using a 3T scanner will be performed for volumetric reconstruction of gray matter on the first 60 participants in both the patient and research volunteer groups. In addition, high-resolution MRI using 7T scanner will be obtained to identify focal structural differences on individual basis in the same 20 SD patients compared to 20 controls. DTI will be conducted for visualization of white matter tracts in 25 subjects per group. The remaining subjects will only undergo the screening and anatomical MRI scans prior to brain donation.

In the postmortem phase, the study will employ MRI of the postmortem brain specimens for diagnostic purposes. Brain and laryngeal tissue will be processed histologically to quantify morphological abnormalities between the two groups. Because it is estimated that about 48% of subjects who participate in the main MRI study will also grant consent for brain/larynx donation, maximum of additional 30 subjects per group are to be recruited for the study. Many of the previous patients who have participated in Laryngeal and Speech Section protocols in the past will be contacted to determine if they would be interested in participating.

OUTCOME MEASURES:

1. Premortem imaging techniques will determine if there are differences in the brain anatomy of patients with SD compared to MTD, VT and to research volunteers:

   1. Volumetric reconstruction of gray matter regions involved in voice production;
   2. Visualization of the white matter tracts between brain regions of interest.
2. Postmortem MRI will identify discrepancies between premortem and postmortem brains of the same persons with SD in comparisons to MTD, VT and to research volunteers.
3. Microscopic examination of brain sections will determine whether abnormalities can be found in the cortical and subcortical regions involved in voice production in persons with SD that differ from patients with MTD and VT.
4. Microscopic examination of the larynx will determine distribution of motor and sensory nerve endings in persons with SD and in patients with MTD and VT and controls.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy research volunteers and patients with SD, MTD, and VT from 21 years of age will be eligible for the study.

SD PATIENTS:

* A diagnosis of adductor or abductor SD will be based on voice testing and fiberoptic nasolaryngoscopy conducted during the initial interview by an otolaryngologist and speech-language pathologist according to following criteria:

  1. Intermittent strained hoarseness, uncontrolled voice breaks or changes in pitch during vowels, liquids (r & l), semivowels (w & y), during speech are present in adductor SD, or
  2. Prolonged voiceless consonants producing breathy breaks are present in abductor SD,
  3. Less prominent symptoms during whisper, singing or falsetto,
  4. Normal voice and vocal fold movement for protective and emotional laryngeal function, such as cough, laugh or cry.
* Postmortem brain and larynx tissue from SD patients deceased from other than neurological, psychiatric, laryngological causes which would not affect our study as determined by medical history.

MTD PATIENTS:

* Increased phonatory muscle tension in the paralaryngeal and suprahyoid muscles on palpation;
* A consistent hypertonic laryngeal posture for phonation, such as either an anterior-posterior squeeze (pin-hole posture) or ventricular hyperadduction and an absence of SD or vocal tremor as determined by a Speech-Language Pathologist and the staff otolaryngologist;
* Exclusion of other laryngeal pathologies based on a fiberoptic nasolaryngoscopic examination conducted during the initial interview by the staff otolaryngologist.

VT PATIENTS:

* Vocal tremor during vocalization that primarily involves laryngeal structures;
* Exclusion of other laryngeal pathologies based on a fiberoptic nasolaryngoscopic examination conducted during the initial interview by the staff otolaryngologist.

CONTROLS:

* Normal vocal function refers to normal voice quality with a negative history of voice or laryngeal disorders.
* Research volunteers without neurological, psychiatric, otolaryngological problems as determined by medical history and examination by a physician.

EXCLUSION CRITERIA:

* Pregnant women will be excluded from the study until a time when they are no longer pregnant.
* Any individual with a medical history or postmortem diagnoses of one or more of the following contraindications will be excluded from the study:

SD, MTD, AND VT PATIENTS:

* Other laryngeal pathologies as determined by medical history and fiberoptic nasolaryngoscopic examination conducted during the initial screening by the otolaryngologist and speech-language pathologist, such as:

  1. Vocal fold paralysis, paresis, joint abnormality, or neoplasm;
  2. Vocal fold nodules, polyps, carcinoma, cysts, contact ulcers, or chronic laryngitis;
  3. Swallowing problems; airway obstruction
* Speech problems as determined by medical history and examination by the otolaryngologist and speech-language pathologist.
* Neurological diseases and disorders such as stroke affecting the brain regions of interest, movement disorders (e.g., Huntington disease, chorea, myoclonus, Gilles de la Tourette syndrome, Parkinson's disease, progressive supranuclear palsy, and neuroleptic-induced syndromes), brain tumors, traumatic brain injury with loss of consciousness, genetic diseases of the CNS, chronic infections of the nervous system, ataxias, myopathies, myasthenia gravis, demyelinating diseases, epilepsy, alcoholism, and drug dependence.
* Psychiatric diseases and disorders such as schizophrenia, major and/or bipolar depression, and obsessive-compulsive disorder.

CONTROLS:

* Laryngeal pathologies as determined by medical history and fiberoptic nasolaryngoscopic examination conducted during the initial screening by the otolaryngologist and speech-language pathologist, such as:

  1. Spasmodic dysphonia, muscular tension dysphonia, voice tremor;
  2. Vocal fold paralysis, paresis, joint abnormality, or neoplasm;
  3. Vocal fold nodules, polyps, carcinoma, cysts, contact ulcers, or chronic laryngitis;
  4. Swallowing problems;
* Speech problems as determined by medical history and examination by the otolaryngologist and a speech-language pathologist.
* Neurological diseases and disorders such as stroke affecting the brain regions of interest, movement disorders (e.g., Huntington disease, chorea, myoclonus, Gilles de la Tourette syndrome, essential tremor, Parkinson's disease, progressive supranuclear palsy, and neuroleptic-induced syndromes), tumors involving the brain region of interest, genetic diseases of the CNS, traumatic brain injury with loss of consciousness chronic infections of the nervous system, ataxias, myopathies, myasthenia gravis, demyelinating diseases, epilepsy, alcoholism, and drug dependence.
* Psychiatric diseases and disorders such as schizophrenia, major and/or bipolar depression, and obsessive-compulsive disorder.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2005-07-14 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Premortem imaging techniques will determine if there are differences in the brain anatomy of patients with SD compared to MTD, VT andto research volunteers | on going
  Premortem imaging techniques will determine if there are differences in the brain anatomy of patients with SD compared to MTD, VT and to research volunteers:a) Volumetric reconstruction of gray matter regions involved in voice production;b) Visualization of the white matter tracts between brain regions of interest.
Postmortem MRI will identify discrepancies between premortem and postmortem brains of the same persons with SD in comparisons to MTD, VT and to research volunteers | after postmortem MRI
  Postmortem MRI will identify discrepancies between premortem and postmortem brains of the same persons with SD in comparisons to MTD, VT and to research volunteers
Microscopic examination of brain sections will determine whether abnormalities can be found in the cortical and subcortical regions involved in voice production in persons with SD that differ from patients with MTD and VT | Postmortem
  Microscopic examination of brain sections will determine whether abnormalities can be found in the cortical and subcortical regions involved in voice production in persons with SD that differ from patients with MTD and VT
Microscopic examination of the larynx will determine distribution of motor and sensory nerve endings in persons with SD and in patients with MTD and VT and controls | Postmortem
  Microscopic examination of the larynx will determine distribution of motor and sensory nerve endings in persons with SD and in patients with MTD and VT and controls

CONTACTS AND LOCATIONS:
Overall Officials: Sandra B Martin, Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Altschuler SM, Bao XM, Bieger D, Hopkins DA, Miselis RR. Viscerotopic representation of the upper alimentary tract in the rat: sensory ganglia and nuclei of the solitary and spinal trigeminal tracts. J Comp Neurol. 1989 May 8;283(2):248-68. doi: 10.1002/cne.902830207. PMID 2738198
- [Background] Aminoff MJ, Dedo HH, Izdebski K. Clinical aspects of spasmodic dysphonia. J Neurol Neurosurg Psychiatry. 1978 Apr;41(4):361-5. doi: 10.1136/jnnp.41.4.361. PMID 650244
- [Background] Aronson AE, Lagerlund TD. Neuroimaging studies do not prove the existence of brain abnormalities in spastic (spasmodic) dysphonia. J Speech Hear Res. 1991 Aug;34(4):801-11. doi: 10.1044/jshr.3404.801. No abstract available. PMID 1956188
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2005-N-0189.html